CLINICAL TRIAL: NCT07174973
Title: Innovative Approaches to Enhance Balance and Neuroplasticity in Multiple Sclerosis: Evaluating the Combined Effects of Transcutaneous Spinal Cord Stimulation, Functional Electrical Stimulation, and Visual Feedback Balance Training
Brief Title: Innovative Approaches to Enhance Balance and Neuroplasticity in Multiple Sclerosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Direct MS Canada (Unknown)
Responsible Party: Principal Investigator, Kei Masani, Principal Investigator, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1431505
Record Dates: First submitted 2025-08-01; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis; Mobility Limitation; Balance; Distorted; Gait
Keywords: balance; neuromodulation; neuroplasticity; multiple sclerosis; mobility
MeSH Terms: conditions — Multiple Sclerosis; Mobility Limitation | interventions — proto-oncogene protein c-fes-fps

STUDY DESIGN:
Intervention Model Description: This study is a pilot, assessor-blinded, randomized, sham-controlled trial.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Balance training only (Sham Comparator): Participants in this group complete the standardized balance training program with sham electrical stimulation.
  Interventions: Other: Balance training only
- Balance training with FES (Active Comparator): This group will receive active FES+ sham TSCS (FES only group) duing balance training
  Interventions: Other: Balance training with FES
- Balance training wiith combined neuromodulation (TSCS+FES) (Active Comparator): This group will receive both TSCS & FES (combined neuromodulation) during balance training
  Interventions: Other: Balance training wiith combined neuromodulation (TSCS+FES)

INTERVENTIONS:
Other: Balance training with FES — Participants assigned to this group complete a standardized balance training program while receiving FES to the lower limb muscles. Training sessions involve standing in a safety harness and performing interactive, game-based balance tasks on a force plate that provides real-time visual feedback of body sway.
  FES will be applied bilaterally to specific leg muscles (e.g., tibialis anterior, quadriceps, gastrocnemius) using surface electrodes. Stimulation parameters (pulse width, frequency, and amplitude) are individually adjusted to produce visible yet comfortable muscle contractions that support functional standing and balance activities. Stimulation is delivered in synchrony with balance exercises to augment muscle activation during postural adjustments.
  Arms: Balance training with FES
Other: Balance training wiith combined neuromodulation (TSCS+FES) — Participants in this group complete the standardized balance training program while receiving both FES and TSCS. Training sessions take place in a safety harness and involve interactive, game-based balance exercises performed on a force plate with real-time visual feedback of body sway.FES is delivered bilaterally to lower limb muscles (e.g., tibialis anterior, quadriceps, gastrocnemius) through surface electrodes. Stimulation parameters (pulse width, frequency, amplitude) are individualized to produce visible, comfortable contractions that facilitate muscle activation during postural tasks.TSCS is applied simultaneously via electrodes placed over the thoracolumbar spinal region to modulate spinal excitability and enhance neuromuscular control. Standardized stimulation parameters are used across participants, with adjustments made to ensure tolerance and safety.
  Arms: Balance training wiith combined neuromodulation (TSCS+FES)
Other: Balance training only — Participants in this group complete the standardized balance training program without electrical stimulation. Sessions are conducted in a safety harness and consist of interactive, game-based balance exercises performed on a force plate, which provides real-time visual feedback of body sway. Tasks are designed to challenge postural control by requiring weight shifting in multiple directions, maintaining stability during perturbations, and progressively increasing task difficulty.
  Arms: Balance training only

SUMMARY:
This study will evaluate the effects of combining balance training with electrical stimulation techniques in individuals with Multiple Sclerosis (MS). MS commonly impairs leg strength, coordination, and balance, increasing the risk of falls and reducing independence. The interventions include:Balance training only, Balance training with Functional Electrical Stimulation (FES), and Balance training with FES and Transcutaneous Spinal Cord Stimulation (TSCS). FES delivers small electrical pulses to leg muscles, while TSCS delivers electrical signals through the skin to stimulate the spinal cord and enhance motor control.

The study will enroll up to 24 participants over a 3-year period. This trial is funded by MS Canada. Participants will be randomly assigned to one of three groups: (1) balance training only, (2) balance training with FES, or (3) balance training with FES and TSCS. All participants will complete 12 supervised training sessions over 6 weeks. During each session, participants will engage in interactive balance games while standing in a safety harness.Outcome assessments will be conducted at three time points: baseline (prior to training), post-intervention (after 6 weeks), and follow-up (8 weeks after training).

Assessments will include:

* Clinical tests of mobility and balance (Timed Up and Go:TUG, 10-Meter Walk Test:10MWT, Berg Balance Scale:BBS)
* Computerized balance testing using a force plate
* Questionnaires on walking ability, fear of falling, and balance confidence
* Neurophysiological measures of brain-spinal cord-muscle communication before and after training

ELIGIBILITY:
Participants will be eligible if they meet the following conditions:

* Confirmed diagnosis of Multiple Sclerosis (MS) according to the revised McDonald criteria
* Age ≤ 65 years
* Ability to walk at least 100 meters, with or without an assistive device, and without requiring rest
* Self-reported perception of impaired balance during standing or walking in daily activities

Exclusion Criteria:

* Participants will be excluded if they present with any of the following:
* Uncorrected visual problems
* Cognitive impairment affecting comprehension of instructions or completion of self-administered outcome measures
* Ongoing MS exacerbation or paroxysmal vertigo
* Concurrent neurological or orthopedic conditions affecting balance
* Recent participation in rehabilitation therapies (physical therapy, occupational therapy, or vestibular therapy) within one month prior to recruitment
* Planned or recent injection of botulinum toxin to the legs during the intervention period
* Peripheral nerve damage affecting the legs
* Contraindications to electrical stimulation, including:implanted electronic device, active cancer or radiation treatment within the past 6 months, uncontrolled epilepsy, skin rash or open wound at electrode site, pregnancy, active deep vein thrombosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-10-30 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go (TUG) | -Baseline (Week 0, prior to intervention start) -Post-intervention (Week 6, within 1 week after completion of the 12 training sessions) - Follow-up (Week 8 post-intervention, approximately Week 14 from baseline)
  Participants begin seated in a standard chair with their back against the chairrest and arms on the armrests. On the command "go," they stand up, walk 3 meters at a comfortable and safe pace, turn around, return to the chair, and sit down. The time to complete the task is recorded in seconds, with shorter times indicating better mobility. For the dual-task cognitive TUG, participants perform the same procedure while simultaneously completing a cognitive task (counting backward by threes). The score is the time in seconds to complete the task, with shorter times indicating better mobility.
10-Meter Walk Test (10MWT) | -Baseline (Week 0, prior to intervention start) -Post-intervention (Week 6, within 1 week after completion of the 12 training sessions) - Follow-up (Week 8 post-intervention, approximately Week 14 from baseline)
  10MWT is a standardized clinical measure of walking speed. Participants are instructed to walk a distance of 10 meters at their usual comfortable pace.Timing is recorded over the middle 6 meters to eliminate the effects of acceleration and deceleration, with 2-meter lead-in and 2-meter lead-out zones. The test is performed twice, and the average walking speed (meters/second) is calculated with faster speeds indicating better mobility.
Berg Balance Scale (BBS): | -Baseline (Week 0, prior to intervention start) -Post-intervention (Week 6, within 1 week after completion of the 12 training sessions) - Follow-up (Week 8 post-intervention, approximately Week 14 from baseline)
  BBS is a 14-item clinical assessment of static and dynamic balance. Each item evaluates performance on a functional task such as standing unsupported, reaching forward, turning, or standing on one leg. Tasks are scored on a 5-point ordinal scale ranging from 0 (unable to perform) to 4 (independent performance), with a maximum total score of 56. Higher scores indicate better balance
Static & Dynamic balance tests | -Baseline (Week 0, prior to intervention start) -Post-intervention (Week 6, within 1 week after completion of the 12 training sessions) - Follow-up (Week 8 post-intervention, approximately Week 14 from baseline)
  For the static balance test, participants will stand for 100 seconds on a force plate under two conditions: (1) eyes open and (2) eyes closed. For the dynamic balance test, participants will stand on the force plate and lean as far as possible in the forward, backward, and sideways directions. During these tasks, body sway, postural movements will be recorded. Visual feedback of calculated body sway will be displayed on a monitor, and participants will be instructed to shift their body toward the indicated directions.
MS Walking Scale-12 (MSWS-12) | -Baseline (Week 0, prior to intervention start) -Post-intervention (Week 6, within 1 week after completion of the 12 training sessions) - Follow-up (Week 8 post-intervention, approximately Week 14 from baseline)
  MSWS-12 is a self-reported questionnaire that measures the impact of Multiple Sclerosis on walking ability. It consists of 12 items in which participants rate, on a 5-point scale (from 1 = not at all to 5 = extremely), how much MS has affected various aspects of their walking during the past two weeks (e.g., walking distance, running, climbing stairs, balance while walking). Scores are summed, transformed to a 0-100 scale, and higher values indicate greater perceived walking limitation. The MSWS-12 is widely used in MS research and clinical practice and has demonstrated strong reliability and validity.
Falls Efficacy Scale-International (FES-I) | -Baseline (Week 0, prior to intervention start) -Post-intervention (Week 6, within 1 week after completion of the 12 training sessions) - Follow-up (Week 8 post-intervention, approximately Week 14 from baseline)
  FES-I is a self-report questionnaire that assesses concern about falling during everyday activities. It includes 16 items rated on a 4-point scale (1 = not at all concerned to 4 = very concerned), covering a range of indoor and outdoor tasks such as getting dressed, bathing, walking on uneven surfaces, or going out sociall
Activities-Specific Balance Confidence (ABC) Scale | -Baseline (Week 0, prior to intervention start) -Post-intervention (Week 6, within 1 week after completion of the 12 training sessions) - Follow-up (Week 8 post-intervention, approximately Week 14 from baseline)
  ABC Scale is a 16-item self-report questionnaire that measures an individual's confidence in maintaining balance during common daily activities. Participants rate their confidence for each activity (e.g., standing on tiptoes, walking on icy sidewalks, reaching, or using an escalator) on a scale from 0% (no confidence) to 100% (complete confidence).
Technology Acceptance Model (TAM) questionnaire | -Baseline (Week 0, prior to intervention start) -Post-intervention (Week 6, within 1 week after completion of the 12 training sessions) - Follow-up (Week 8 post-intervention, approximately Week 14 from baseline)
  TAM questionnaire is a validated self-report tool used to assess user acceptance of new technologies. It measures key domains including perceived usefulness (the extent to which the technology improves task performance), perceived ease of use (the degree to which the technology is user-friendly), attitudes toward use, and behavioral intention to use. Items are typically rated on a Likert-type scale, and higher scores indicate greater acceptance.

SECONDARY OUTCOMES:
Neurophysiological assessment:corticospinal excitability | -Baseline (Week 0, prior to intervention start) -Post-intervention (Week 6, within 1 week after completion of the 12 training sessions) - Follow-up (Week 8 post-intervention, approximately Week 14 from baseline)
  The strength of the connection between the brain and muscles will be measured using TMS. During this test, the participant sits comfortably in a chair while a small device placed over the head delivers brief magnetic pulses. These pulses activate specific brain areas and the responses in the muscles are recorded, providing information about brain-muscle communication.The MEP (motor evoked potential) score is the amplitude of the muscle response in microvolts (µV or mV), with larger amplitudes indicating stronger corticospinal excitability and smaller or absent responses reflecting weaker or impaired brain-muscle connectivity.

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto Rehabilitation Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No